CLINICAL TRIAL: NCT01999595
Title: The Effect of Pulse Frequency and Pad Size of Transcutaneous Electrical Nerve Stimulation (TENS) on Experimental Blunt Pressure Pain in Healthy Participants
Brief Title: The Antalgic Effect of Pulse Frequency and Pad Size of TENS on Blunt Pressure Pain
Acronym: TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Hung Kaung University (Other)
Responsible Party: Principal Investigator, Chih Chung Chen, Assistant Professor in Department of Physical Therapy, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102-4765B; HK-99-B-07 (Other: Hung Kuang University)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Transcutaneous Electrical Nerve Stimulation; Blunt Pressure Pain; Pad Size; Pulse Frequency; Analgesia
Keywords: transcutaneous electrical nerve stimulation; pad size; pulse frequency; blunt pressure pain; healthy humans.
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: One hundred eighty participants (equal number of females and males, Fig. 1) were randomly assigned into six groups with the following TENS characteristics. (1) Group 1:
  control group, (2) group 2: sham group, (3) group 3: high frequency (80 pps)/large pad (5 cm x 10 cm) group, (4) group 4: low frequency (3 pps)/large pad (5 cm x 10 cm) group, (5) group 5: high frequency (80 pps)/small pad (5 cm x 2.5 cm) group, and (6) group 6: low frequency (3 pps)/small pad (5 cm x 2.5 cm) group.
Who Masked: Participant, Investigator
Masking Description: The group allocation for each participant was sealed in an envelope prepared by an investigator. Just before the start of the second visit, a second investigator opened the envelope to confirm the allocation of TENS groups for individual participants and applied the TENS. For better blinding, a third investigator assessed the blunt pressure pain threshold (BPPT) for the baseline value.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- High frequency TENS with large pads (Experimental): TENS=transcutaneous electrical nerve stimulation
  High frequency TENS was a 80 Hz TENS delivered via a pair of electrodes with the size of 5 cm x 10 cm
  Dosage: same as electrical density using a standardized pad size (5cm x 5cm) with comfortable intensity
  Interventions: Device: High frequency TENS with large pads
- Low frequency TENS with large pads (Experimental): TENS=transcutaneous electrical nerve stimulation
  Low frequency TENS was a 3 Hz TENS delivered via a pair of electrodes with the size of 5 cm x 10 cm
  Dosage: same as electrical density using a standardized pad size (5cm x 5cm) with comfortable intensity
  Interventions: Device: Low frequency TENS with large pads
- High frequency TENS with small pads (Experimental): TENS=transcutaneous electrical nerve stimulation
  High frequency TENS was a 80 Hz TENS delivered via a pair of electrodes with the size of 5 cm x 2.5 cm
  Dosage: same as electrical density using a standardized pad size (5cm x 5cm) with comfortable intensity
  Interventions: Device: High frequency TENS with small pads
- Low frequency TENS with small pads (Experimental): TENS=transcutaneous electrical nerve stimulation
  Low frequency TENS was a 3 Hz TENS delivered via a pair of electrodes with the size of 5 cm x 2.5 cm
  Dosage: same as electrical density using a standardized pad size (5cm x 5cm) with comfortable intensity
  Interventions: Device: Low frequency TENS with small pads
- Control TENS (Placebo Comparator): TENS=transcutaneous electrical nerve stimulation
  Control TENS was the application of electrical stimulation via skin with no current
  Interventions: Device: Control TENS
- Sham TENS (Sham Comparator): TENS=transcutaneous electrical nerve stimulation
  Sham TENS was the application of electrical stimulation via skin with no current on the participant, who was told that the TENS was "turn-on" whether you feel it or not
  Interventions: Device: Sham TENS

INTERVENTIONS:
Device: Control TENS — Control TENS was the application of electrical stimulation via skin with no current
  Arms: Control TENS
Device: Sham TENS — Sham TENS was the application of electrical stimulation via skin with no current on the participant, who was told "TENS is at a turn-on level whether or not you feel it"
  Arms: Sham TENS
Device: High frequency TENS with large pads — High frequency TENS was delivered on large electrodes
  Arms: High frequency TENS with large pads
Device: Low frequency TENS with large pads — Low frequency TENS was delivered on large electrodes
  Arms: Low frequency TENS with large pads
Device: High frequency TENS with small pads — High frequency TENS was delivered on small electrodes
  Arms: High frequency TENS with small pads
Device: Low frequency TENS with small pads — Low frequency TENS was delivered on small electrodes
  Arms: Low frequency TENS with small pads

SUMMARY:
The purpose of this study is to determine the antalgic of surface electrical stimulation with pulse frequencies and pad sizes on blunting pressure pain on healthy human due to various temporal and spatial summations of the stimulation.

DETAILED DESCRIPTION:
Potential participants expressing interest in the study will be given to read the contraindications for the pain tests and the stimulation intervention, which has been documented on the consent form. All participants meeting entry requirements will be invited to participate in the experiments which take place on a separate occasion.

Each participant will sign the consent form and will be told again that they can withdraw from the study at any time and without explanation. Each participant will be required to experience a 10-minute pre-stimulation period, a 30 minute TENS intervention, a 30 minute follow-up period.

Participants will be seated on a chair with arm support provided by a side table. The investigator will be then informed the stimulation intervention and used pad size on the stimulation periods in written form contained in a sealed envelope. After the participant's verbal permission is obtained, the investigator will apply the pads on the dorsal forearm area.

Either the large size pad, 5cm x 10cm, or the small size,2.5cm x 2.5cm, will be choose to place on the dorsal side of the forearm to straddle the site for blunt pressure pain. The muscle bellies of the forearm are mainly located on the proximal half part. The proximal pad will be attached to the lateral epi-condyle of the elbow, and the distal electrode will be placed 3cm distal to the proximal one along the line between the lateral part of elbow and the mid-point of the wrist. The pads will be then connected to the intervention stimulator. The investigator will relay instructions to the participants using cue cards displayed 30 seconds before any required action.

Before each blunting pressure pain test, the participant will sit comfortably and place their right upper extremity on a side table with the shoulder abduction, elbow flexion, the forearm pronation. The test will be induced using a pressure algometer with a flat circular probe, measuring 1.1cm in diameter (1cm2 on skin surface). Force will be displayed digitally in increments of 0.1 Newton. The algometer will be applied to the mid-point between the intervention pads. The rate of the pressure algometer application will be around 6 Newtons per second on average. The participants will be asked to concentrate on the sensations in the forearm. When the pressure becomes definitely painful, the participant will state "Pain!" and the force will be stopped. The pain threshold will be taken twice in a minute for one test and each measurement will take no more than 30 seconds.

There will be seven 1-minute tests performed in this experiment. The first test in pre-stimulation period. The second and third tests were administered and started at 9, 19, 29 minute time points in the stimulation-on period. A 30 minute post stimulation period will be then followed. Another 3 tests will be performed in this period in ten-minute intervals at 39, 49, 59 minute time points after the stimulation start.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and aged 18 years or over

Exclusion Criteria:

* Any open wound around the arm or hand area, including edema or inflammation;
* Cardiac or vascular problems (such as coronary artery disease, coronary thrombosis, or angina pain, high blood pressures, phlebitis, and pacemaker implantation);
* Any dermatological problems or infections around the hand, forearm, or arm area (such as dermatitis or eczema, bacterial or fungal infections);
* Any history of neoplasm or malignancy;
* Bleeding diseases on the arm or hand (such as haemorrhage); Menstruation or pregnancy;
* Abnormal neurological signs in the upper limbs (such as altered skin sensations);
* Hypersensitivity or phobia to electrical application;
* Any current medication regime.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2013-05-30 (Actual); Study Completion 2013-05-30 (Actual)

PRIMARY OUTCOMES:
blunting pressure pain threshold | 6 months
  The test will be induced using a pressure algometer with a flat circular probe, measuring 1.1cm in diameter (1cm2 on skin surface). Force will be displayed digitally in increments of 0.1 Newton. The algometer will be applied to the mid-point between the electrodes. The rate of the pressure algometer application will be around 6 Newtons per second on average. The participants will be asked to concentrate on the sensations in the forearm. When the pressure becomes definitely painful, the participant will state "Pain!" to stop the pressure force.

CONTACTS AND LOCATIONS:
Overall Officials: Chih Chung Chen, D.Ph., Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Guishan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chesterton LS, Foster NE, Wright CC, Baxter GD, Barlas P. Effects of TENS frequency, intensity and stimulation site parameter manipulation on pressure pain thresholds in healthy human subjects. Pain. 2003 Nov;106(1-2):73-80. doi: 10.1016/s0304-3959(03)00292-6. PMID 14581113
- [Result] Chesterton LS, Barlas P, Foster NE, Baxter DG, Wright CC. Gender differences in pressure pain threshold in healthy humans. Pain. 2003 Feb;101(3):259-266. doi: 10.1016/S0304-3959(02)00330-5. PMID 12583868
- [Result] Chesterton LS, Barlas P, Foster NE, Lundeberg T, Wright CC, Baxter GD. Sensory stimulation (TENS): effects of parameter manipulation on mechanical pain thresholds in healthy human subjects. Pain. 2002 Sep;99(1-2):253-62. doi: 10.1016/s0304-3959(02)00118-5. PMID 12237203